CLINICAL TRIAL: NCT01525277
Title: The Side of Implantable Central Vascular Catheters and Complications in Cancer Patients: A Randomization Observational Study
Brief Title: The Side of Implantable Central Vascular Catheters and Complications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201110050RB
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Upper Extremity Deep Vein Thrombosis, Secondary
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- left subclavian vein: CVC implanted in the left subclavian vein
- right subclavian vein: CVC implanted in the right subclavian vein

SUMMARY:
Whether the side of implantable CVCs was associated with the complication rates remains unclear. The investigators plan this study to explore this issue by randomizing patients to receive CVC implantation at the left subclavian or righ subclavian vein.

DETAILED DESCRIPTION:
Implantable central venous catheters (CVC) are crucial for cancer patients. They provide central venous access for chemotherapy and high-concentration nutrition support. However, several potential CVC-related complications may develop and severely interfere with the patients' cancer treatment and can be life-threatening in some occasions.

Thrombotic events occurred in around 20% of cancer patients with implantable CVCs. Such events included intraluminal thrombosis and catheter-related venous thrombosis. Catheter removal was usually necessary to resolve these conditions. Treatment delays are inevitable for these patients. Besides, these thrombotic complications were associated with catheter-related infection, which could be highly dangerous for cancer patients.

Risk factors associated with these thrombotic events included the hypercoagulable state of the patients, the cancer types, the catheter types, and the placement of the catheter tips in the superior vena cava. Some single-arm studies found that CVC inserted from the left subclavian veins led to more CVC-related thrombosis than those inserted from the right subclavian vein. However, for most right-handed patients, to place these implantable CVCs on the right side is inconvenient for daily life because vigorous exercise was then impossible. Besides, these single-arm studies could not well control the other potentially interfering factors, such as the operators, catheter location and cancer types.

Therefore, we plan a randomized observational study to explore whether the side of implantable CVCs was actually associated with the complication rates. Cancer patients who need implantable CVCs will be randomized to have the catheters implanted either in the left subclavian vein or the right subclavian. Patients who had breast cancer, mediastinal mass with the diameter > 6 cm, ECOG performance score >2, or those who were not able to receive a standing P-A view chest X-ray will be excluded. Patients who had other reasons that prevented the randomization will also be excluded. The catheter-related complications will be actively reported by the patients. We will also enforce the records of complications by chart reviews and regular telephone contacts.

With the study, we can demonstrate whether a left-sided CVC and a right-sided CVC are different in complication rates. The result should be very useful in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients who required implantable CVCs
2. Age > 20
3. Not previously implanted with implantable CVCs in subclavian veins.

Exclusion Criteria:

1. Breast cancer patients
2. Mediastinal mass > 6 cm
3. ECOG performance score > 2
4. Not able to receive a standing P-A view chest X-ray exam.
5. One of the subclavian veins has problems preventing randomization

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients who required implantable CVCs
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
complication rates | everey 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Yun Shao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan